CLINICAL TRIAL: NCT00948350
Title: Anesthesia for Awake Fiberoptic Intubation in Patients With Cervical Instability - Comparison of Translaryngeal Injection and "Spray as You go"-Technique
Brief Title: Anesthesia for Awake Fiberoptic Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinikum St. Georg gGmbH (Other)
Responsible Party: Principal Investigator, Armin Sablotzki, MD, Prof. Dr. med., Klinikum St. Georg gGmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EK-BR-34/08-1; Stu08/0041
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Intubation
Keywords: cervical instability; awake intubation; laryngeal anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- translaryngeal injection (Active Comparator): translaryngeal injection of local anesthetics before the awake intubation
  Interventions: Procedure: awake intubation
- spray as you go (Active Comparator): local anesthetics are given through the fiberoptic during awake intubation
  Interventions: Procedure: awake intubation

INTERVENTIONS:
Procedure: awake intubation — two anesthesia techniques

SUMMARY:
This is a prospective, comparative, randomized, monocentric, clinical open study, to compare two anesthesia techniques (translaryngeal injection vs. spray as you go) in patients with cervical instability with regard to technical modalities and quality of fiberoptic awake intubation.

DETAILED DESCRIPTION:
In patients with cervical instability anesthesia induction and conventional intubation are associated with the risk of neurological harm. Therefore the method of choice for anesthesia induction is the fiberoptic awake intubation. This method allows to place the ventilation tube without movement of the cervical spinal cord. This procedure is very uncomfortable for the patient and needs the application of topic and/or systemic anesthetics.

With this clinical study we will compare two established techniques for local laryngeal anesthesia with regard to the quality of technical modalities and postoperative outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients with cervical instability undergoing elective decompression of cervical spine

Exclusion Criteria:

* patient refused participation
* contraindications for awake intubation techniques (e.g. nasal bleeding, anatomical disorders)
* patient under alcohol or drugs
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
patients satisfaction with anesthesia | up to two weeks after hospital admission
  participants will be followed for the duration of hospital stay, an expected average of 2 weeks

SECONDARY OUTCOMES:
pain after anesthesia | Change from Baseline in pain after anesthesia at end of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Armin R Sablotzki, MD, Study Chair — Clinics of Anesthesiology, Critical care and Pain Therapy; Michael Malcharek, MD, Principal Investigator — Clinic of Anesthesiology, Dept. Neuroanesthesia and Neuromonitoring
Locations (1):
- Klinikum St. Georg gGmbH, Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Malcharek MJ, Bartz M, Rogos B, Gunther L, Sablotzki A, Gille J, Schneider G. Comparison of Enk Fibreoptic Atomizer with translaryngeal injection for topical anaesthesia for awake fibreoptic intubation in patients at risk of secondary cervical injury: A randomised controlled trial. Eur J Anaesthesiol. 2015 Sep;32(9):615-23. doi: 10.1097/EJA.0000000000000285. PMID 26086284